CLINICAL TRIAL: NCT05022602
Title: Clinical Evaluation of Opto-Acoustic Image Quality With the Gen 2 Imagio System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seno Medical Instruments Inc. (Industry)
Collaborators: American College of Radiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Gen 2 - 01
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Imagio (Experimental): Imagio Grayscale only probe and Imagio Duplex probe in ultrasound only and OA modes
  Interventions: Device: Imagio

INTERVENTIONS:
Device: Imagio — Imagio - both ultrasound probe and Duplex OA probe

SUMMARY:
This study performs the first clinical evaluation of the Gen 2 Imagio System in a clinical setting to assess image quality with both the IUS ultrasound only probe and the OA/US (duplex probe).

DETAILED DESCRIPTION:
1. Obtain ultrasound only probe images and duplex probe OA/US (both gray scale and OA) probe images. This includes doppler and elastography imaging with the gray scale only ultrasound probe and ultrasound mode of the duplex OA/US probe.
2. Provide breast and lymph node pathology results (except BI-RADS 1, 2 and 3 (as applicable))

ELIGIBILITY:
Inclusion Criteria:

1. Has a signed and dated informed consent, prior to initiation of any study-related activities.
2. Is at least 18 years of age.
3. Have been referred for a breast US because of a breast lesion/mass finding via a palpable lump or per standard of care imaging.
4. Is willing and able to comply with protocol-required scans

Exclusion Criteria:

1. Is pregnant or lactating.
2. Has a condition or breast impediment (i.e. insect bites, poison ivy, rash, open wounds, chafing of the skin, scar, tattoos, moles, hematoma, nipple rings, etc.) which could interfere with the intended field of view.
3. Is experiencing photo-toxicity associated with currently taking, or having taken, photosensitizing agents within the previous 72 hours such as some sulfur containing drugs, ampicillin, tetracycline.
4. Is currently undergoing phototherapy.
5. Has a history of any photosensitive disease (e.g., porphyria, lupus erythematosus) or undergoing treatment for a photosensitive disease and is experiencing photosensitivity.
6. Has had an adverse reaction in the past to medical laser procedures, such as laser hair removal or laser tattoo removal.
7. Has had prior benign excisional breast biopsy on breast of interest within the past 18 months.
8. Currently has mastitis.
9. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pam Otto, MD, Principal Investigator — UTHSC
Locations (1):
- UT Health, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imagio
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imagio
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (15.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Imagio Image Sets Collected
Description: Obtain ultrasound only probe images and OA/US (both gray scale and OA) probe images as measured by the receipt of image sets for each subject enrolled.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Imagio
Number analyzed (Participants) | 38
Participants | 38

2. Primary Outcome: Number of Subjects With Completed Pathology Results
Description: Provide breast pathology results per subject (except BI-RADS 1, 2 and 3 (as applicable)) if subject's study mass is biopsied
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Imagio
Number analyzed (Participants) | 38
Participants | 23

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time the patient entered the Imagio imaging room until they departed from the facility the same day. There were no follow-up exams for this study (up to 3 hours).
Arm/Group | Imagio
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 1/38
OTHER ADVERSE EVENTS (reported when occurring in more than 2.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imagio (N=38)
Medical Device Site Warmth (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INSTITUTION/INVESTIGATOR will provide such proposed publications/presentations, to SPONSOR for review, at least thirty (30) days prior to submission for publication or of public disclosure. SPONSOR will complete its review within thirty (30) days of receipt of the submitted publications/presentations. The INSTITUTION shall consider SPONSOR's suggestions and comments to the manuscript to be published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT05022602/Prot_SAP_000.pdf